CLINICAL TRIAL: NCT02325817
Title: A Multicenter, Superior, Randomized Controlled Clinical Trial to Observe the Safety and Efficacy of Bingo Drug-eluting Balloon vs. Yinyi Balloon Dilatation Catheter in the Treatment of Patients With Bifurcation Stenosis Lesions of Coronary Artery
Brief Title: Bingo Drug-eluting Balloon in Bifurcation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yinyi(Liaoning) Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEYOND
Record Dates: First submitted 2014-12-20; First posted 2014-12-25 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Bifurcation Lesions; Drug Eluting Balloon
Keywords: Bifurcation Lesions; drug eluting balloon; paclitaxel; drug coated balloon

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug-eluting balloon (Experimental): Treat the side branch of bifurcation lesion with drug-eluting balloon
  Interventions: Device: Drug-eluting balloon
- Uncoated balloon (Active Comparator): Treat the side branch of bifurcation lesion with uncoated balloon
  Interventions: Device: Uncoated ballloon

INTERVENTIONS:
Device: Drug-eluting balloon — Treat the side branch of bifurcation lesion with drug-eluting balloon
  Arms: Drug-eluting balloon
Device: Uncoated ballloon — Treat the side branch of bifurcation lesion with uncoated balloon
  Arms: Uncoated balloon

SUMMARY:
The purpose is to observe and evaluate the safety and efficacy of Bingo drug-eluting balloon in the treatment of patients with bifurcation lesions of coronary artery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female ages 18-80 years old
2. Patients with asymptomatic myocardial ischemia symptom, stable or unstable angina pectoris or old myocardial infarction
3. Patients with bifurcation lesions of coronary artery observed by angiography.
4. The main branch of the vessels are suitable for PCI and stent therapy, and the side branch are intended to implement the kissing dilatation without considering dual stent implantation.
5. De Novo bifurcation lesions and diameter stenosis are not less than70%;
6. Referenced vessel diameters range from 1.25mm to 5.0mm, and lesions range are not more than 40mm
7. Residual stenosis are not more than 50% after predilatation;
8. Patients who understand the purpose of this trial, voluntary and sign informed consent.

Exclusion Criteria:

1. Heavily calcified lesions which cannot be dalatated successfully, and the lesions which are not suitable by balloon angioplasty
2. Left main coronary artery lesions without protection or related bifurcation lesions
3. Patients with severe heart failure symptoms (above NYHA III) or Left ventricular ejection fraction (LVEF) below 35% (ultrasound or left ventricular angiography)
4. Impairment of the renal function preoperative: Serum creatinine above 2.0mg/dl；
5. Patients with hemorrhagic tendency, the history of active digestive ulcers, the history of subarachnoid hemorrhage cerebral hemorrhage, antiplatelet and anticoagulant therapy contraindication and unable to anticoagulant therapy;
6. Patients who are allergic to aspirin, ticagrelor, clopidogrel, ticlopidine, heparin, contrast agent and paclitaxel, and cannot 1-year tolerate dual antiplatelet therapy (aspirin + clopidogrel or ticagrelor)
7. Patients whose expected lives are less than 1 year;
8. Patients who are considered to have poor compliance and cannot complete the trial in accordance with requirements.
9. In-stent restenosis lesions
10. Patients who are enrolled in this trial and need stent therapy due to vascular laceration or severe stenosis, and those patients are calculated as fall off cases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2014-12-03 (Actual); Primary Completion 2016-11-29 (Actual); Study Completion 2017-01-13 (Actual)

PRIMARY OUTCOMES:
Target lesion Stenosis (diameter, %) | 9 months

SECONDARY OUTCOMES:
TLR | 1, 6 and 9 months
TVR | 1, 6 and 9 months
TLF | 1, 6 and 9 months
  cardiac death, target vessel MI, TLR
MACCE | 1, 6 and 9 months
  all-cause death, MI, stroke and TVR
All-cause death | 1, 6 and 9 months
Cardiac death | 1, 6 and 9 months
Non-fatal MI, thrombosis | 1, 6 and 9 months
Thrombosis | 1, 6 and 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Shenyang Military Region, Shenyang, Liaoning, China

REFERENCES:
- [Derived] Jing QM, Zhao X, Han YL, Gao LL, Zheng Y, Li ZQ, Yang P, Cong HL, Gao CY, Jiang TM, Li H, Li JX, Wang DM, Wang G, Cong ZC, Zhang Z. A drug-eluting Balloon for the trEatment of coronarY bifurcatiON lesions in the side branch: a prospective multicenter ranDomized (BEYOND) clinical trial in China. Chin Med J (Engl). 2020 Apr 20;133(8):899-908. doi: 10.1097/CM9.0000000000000743. PMID 32265425